CLINICAL TRIAL: NCT01600404
Title: Effects of Antimuscarinic Drugs on the Cognition of Patients With Acute Spinal Cord Injury
Brief Title: Effects of Antimuscarinics on Cognition in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2011-25
Record Dates: First submitted 2012-05-10; First posted 2012-05-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Mild Cognitive Impairment; Spinal Cord Injuries
Keywords: Mild Cognitive Impairment; Muscarinic Antagonists; Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive; Overactive Detrusor
MeSH Terms: conditions — Cognitive Dysfunction; Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- antimuscarinic treatment: antimuscarinic treatment
  Interventions: Drug: antimuscarinic treatment
- no antimuscarinic treatment (control)

INTERVENTIONS:
Drug: antimuscarinic treatment
  Groups: antimuscarinic treatment

SUMMARY:
Prospective evaluation of the cognitive function of in-house patients suffering from an acute traumatic spinal cord injury before and three months after the initiation of antimuscarinic treatment.

The following hypothesis will be tested: Antimuscarinic treatment results in significantly worse cognitive test results three months after traumatic spinal cord injury compared to the pre-treatment results and the results of the control group.

DETAILED DESCRIPTION:
There will be two groups: 1) patients receiving antimuscarinic treatment 2) patients without antimuscarinic treatment (control).

The control group will be investigated in order to determine the effects of traumatic spinal cord injury on cognition and the natural history of potential cognitive impairment within the first three months after spinal cord injury.

Six to eight weeks after traumatic spinal cord injury, patients are examined in order to determine the type of neurogenic bladder dysfunction they are suffering from. Patients suffering from an overactive bladder will receive antimuscarinic treatment in order to prevent high urine storage and voiding pressures, that put the kidneys at risk.

Prior to the urologic examination, patients fulfilling inclusion criteria will be contacted. If informed consent is given, cognitive function will be evaluated in both patient groups using different standard neuropsychologic tests. The same neuropsychologic tests will be repeated three months later. Evaluation will take place under standardized conditions (e.g. time of day).

Furthermore,different factors influencing cognition, e.g. depression, pain, medication, will be assessed at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* acute traumatic spinal cord injury
* primary rehabilitation / in-house patient
* 18-65 years of age
* treatment group: indication for antimuscarinic treatment (oxybutynin, tolterodine
* willingness and motivation to participate in study

Exclusion Criteria:

* lesion level above C4
* traumatic brain injury (initial Glasgow Coma Score < 13)
* pre-existing dementia
* pre-existing impaired cognitive function
* previous antimuscarinic treatment
* treatment group: antimuscarinic treatment other than oxybutynin, tolterodine
* acute psychologic disorders, diseases, schizophrenia
* alcohol abuse, consumption of illegal drugs (incl. marijuana)
* moderate to severe depression (Beck Depression Inventory Score > 18)
* moderate to severe pain (International Spinal Cord Injury Pain Basic Data Set)
* progressive disease
* tricyclic antidepressant
* color blindness, impaired sight, blindness
* insufficient German language skills
* no informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute (4-8 week post-injury) traumatic spinal cord injury during first rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
d2 Test | change from enrollement to 3 months

SECONDARY OUTCOMES:
International Spinal Cord Injury Pain Basic Data Set | day 0 and at 3 months
Beck Depression Inventory Score | day 0 and at 3 months
patient characteristics | day 0
  age
type of neurologic lower urinary tract dysfunction | day 0
Stroop Test | day 0 and at 3 months
California Verbal Learning Test | day 0 and at 3 months
Verbal Fluency Test according to Thurstone | day 0 and at 3 months
visuospatial performance | day 0 and at 3 months
  subtests from Wechsler Adult Intelligence Scale
divided attention | day 0 and at 3 months
  subtests from test battery according to Zimmermann and Fimm
patient characteristics | day 0
  sex
patient characteristics | day 0
  date of injury
patient characteristics | day 0
  tpe of accident
patient characteristics | day 0
  Glasgow Coma Scale
patient characteristics | day 0
  lesion level
patient characteristics | day 0
  completeness of injury
patient characteristics | day 0
  ASIA impairment score

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, Prof, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland